CLINICAL TRIAL: NCT00934258
Title: Effect of Genes on Rosuvastatin Therapy for Hyperlipidemia
Status: Available | Type: Expanded Access
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200812111R; 200812111R
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Hyperlipidemia
Keywords: genes; rosuvastatin; fenofibrate; Cardiovascular (CV) diseases; dyslipidemia; metabolic syndrome; identify genetic determinants of the wide range of interindividual variability in phenotypic and clinical response to the lipid-lowering drug classes; identify genetic susceptibility to drug-related side effects.
MeSH Terms: conditions — Hyperlipidemias; Disease; Dyslipidemias; Metabolic Syndrome | interventions — Rosuvastatin Calcium; Fenofibrate; Cytochrome P-450 CYP2C9; UDP-Glucuronosyltransferase 1A9

INTERVENTIONS:
Drug: rosuvastatin,fenofibrate — Rosuvastatin 10 mg once daily Rosuvastatin 5 mg + SFC fenofibrate 80 mg
Genetic: CYP2C9, UGT1A1, UGT1A3, OATP2, BCRP — All potential patients will be screened for the eligibility in a screening visit. Those who fill the inclusion criteria at screening will be invited for the registry study into different groups. The follow-up will take place at months 6, 12, 18, and every year thereafter for another 3 years, through clinical visiting, phone follow-up, or records from the NHIB Taiwan. At each clinical visit, vital signs, clinical endpoints, adverse events, concurrent medication information and laboratory specimens will be obtained as complete as possible. With phone or records from NHIB, only clinical endpoints will be recorded. If the primary care physician intends to treat the patient's lipid profile to the target, he/she can add, delete or adjust the LLT by his/her clinical judgement

SUMMARY:
Previous studies indicate that the variant status of detoxification proteins is different among Taiwanese and other ethnic groups. For example, in Taiwanese, the major SNPs of CYP2C9 are CYP2C9*2 (430C>T) and CYP2C9*3 (1075A>C) and their frequencies are different from that in Caucasians [11]. The second example is that the frequency of the A(TA)7TAA allele in the promoter area of the UGT1A1 gene is substantially lower, while for the rate of variation within the coding region is much higher in Taiwanese than that in Caucasians (14.3% vs. 35.7- 41.5% and 29.3% vs. 0.1%, respectively) [12]. The third example is that the frequency of 388A>G of the OATP2 gene in Taiwanese (0.68) [13] is in between that in European Americans (0.30) and African Americans (0.74) [14]. Therefore, the investigators hypothesize that, in Taiwanese the SNPs of detoxification proteins modulate the lipid-lowing effects of RVA and fenofibrate may be different from those for Caucasians.

DETAILED DESCRIPTION:
Since April 2008, we have started to run a multicenter, prospective, randomized, open-label, blinded end-point classification trial to test the hypothesis in Taiwan that the addition of fibrate on statin would provide a further reduction in the major coronary events in the patients with diabetes or atherosclerotic vascular diseases with metabolic syndrome. With the advantage of this large-scaled prospective trial, it is also a good opportunity to identify simultaneously the genetic determinants of wide range of interindividual variability in phenotypic and clinical response to two major lipid-lowering drug classes, rosuvastatin and fenofibrate. The aim of this proposal is to find which SNPs influence the therapeutic effectiveness of lipid lowering therapy in Taiwanese hyperlipidemic patients. A key feature is the use of multiple drug-treated population samples to get the findings derived from both candidate gene and genome-wide searches for SNP associations with markers of drug efficacy as well as side effects. Thus the promise of pharmacogenomics and metabolomics-- "individualized medicine" will come true in treating hyperlipidemia in Taiwanese.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 20-79 years with definite DM or atherosclerotic vascular diseases with metabolic syndrome, defined as the presence of three or more of the following risk factors:

  * abdominal obesity (waist circumference > 90 cm in men or > 80 cm in women),
  * triglycerides > 150 mg/dL, HDL-cholesterol < 40 mg/dL in men or < 50 mg/dL in women,
  * blood pressure > 130/85 mm Hg, or
  * fasting glucose > 100 mg/dL).
* Those who are qualified for lipid lowering therapy according to the Taiwanese national guidelines (LDL-C 130-190 mg/dL or TG 200-500 mg/dL with HDL-C < 40 mg/dL or TC/HDL-C > 5).

Exclusion Criteria:

* Any known contraindications to statin or fibrate therapy,
* Previous intolerance to statin or fibrate in low or high doses,
* Liver enzyme levels more than 3 times the upper limit of normal,
* Pregnancy or breastfeeding,
* Nephrotic syndrome,
* Uncontrolled diabetes mellitus (HbA1c > 9),
* Uncontrolled hypothyroidism,
* Plasma LDL-C level higher than 190 mg/dL or triglyceride level higher than 500 mg/dL,
* Coronary heart disease event or revascularisation within a month,
* Congestive heart failure (New York Heart Association classification IIIb or IV),
* Hemodynamically important valvular heart disease,
* Gastrointestinal conditions affecting absorption of drugs,
* Treatment with other drugs that seriously affect the pharmacokinetics of statins or fibrate,
* Unexplained creatine phosphokinase concentrations six or more times the upper limit of normal,
* Life-threatening malignancy,
* Treatment with immuno suppressive or other lipid lowering drugs.
* Patients previously treated with monotherapy with statins or fibrates will be qualified if they have not already had titration to a dose higher than the equivalent of 5 mg/d of rosuvastatin or 160 mg/d of SFC fenofibrate.

Ages: 20 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult